CLINICAL TRIAL: NCT04568668
Title: Implementing and Evaluating ActionADE to Transform Medication Safety Among Patients With Adverse Drug Reactions
Brief Title: Evaluating ActionADE in Reducing Adverse Drug Reactions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Health, British Columbia (Other Government); Vancouver Coastal Health (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Corinne Hohl, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H18-01332
Record Dates: First submitted 2020-09-05; First posted 2020-09-29 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Adverse Drug Event; Adverse Drug Reaction
Keywords: Health Information Technology; Patient Safety; Health Systems
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: We will conduct a triple-blind randomized controlled trials. We will enroll consecutive eligible patients presenting to the Emergency Department with an adverse drug event to prescribed outpatient medication. Randomization is implemented in the ActionADE application. Randomization will be equal (1:1) and stratified by site and age (< 80, ≥ 80). A statistician otherwise uninvolved in the study will generate a list of treatment assignments using permuted blocks of varying sizes for each stratum. ActionADE will store the randomization list for each stratum. Once eligibility has been determined, the application will allocate the patient to the next available assignment within the stratum.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study participants, outcomes assessors, and study investigators will be blinded to treatment allocation. Community pharmacists cannot be blinded to the intervention, as we are studying the change in pharmacists' dispensing behavior due to the provision of new adverse drug event information. The information will only appear for patients in the experimental arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADE information transmitted to PharmaNet (Experimental): Patients in the experimental arm will have standardized adverse drug event information documented in ActionADE transmitted to and stored in PharmaNet, British Columbia's medication dispensing database. The adverse drug event information will become visible to any subsequent healthcare provider who accesses the patient's PharmaNet profile. Community pharmacy software will import the adverse drug event information such that community pharmacists can view the adverse drug event information prior to dispensing medications.
  Interventions: Device: ActionADE
- Standard care (ADE information retained locally) (No Intervention): Patients in the control group will have their adverse drug event information recorded in ActionADE, and their information will be retained locally, as is the current standard of care. This means that their adverse drug event information will not be visible to other providers via PharmaNet.

INTERVENTIONS:
Device: ActionADE — ActionADE is a software application that allows healthcare providers to document standardized adverse drug event information in a user-friendly and standardized manner. We integrated ActionADE uni-directionally with PharmaNet, a secure province-wide network that links all pharmacies in British Columbia to a central data system. This allows care providers to pull in demographic information and visualize their patient's medication dispensing history.
  In 2020, we enabled bi-directional integration with PharmaNet allowing clinicians to transmit standardized adverse drug event information back to the PharmaNet database. The three dominant community pharmacy systems in the geographic area of the trial will display the adverse drug event information in their systems, and generate patient-specific medication-level alerts when pharmacists attempt to re-dispense a culprit medication.
  Arms: ADE information transmitted to PharmaNet

SUMMARY:
Repeat exposures to culprit medications are a common cause of preventable adverse drug events. Health information technologies have the potential to reduce repeat adverse drug events by improving information continuity. However, they rarely interoperate to ensure providers can view adverse drug events documented in other systems. The investigators designed ActionADE to enable rapid documentation of adverse drug events, and communication of standardized information across health sectors by integrating ActionADE with legacy systems.

The investigators will leverage ActionADE's implementation to conduct a randomized trial on patients diagnosed with adverse drug reactions in the main trial. This study will take place in Vancouver, British Columbia, Canada.

DETAILED DESCRIPTION:
Medication use is rising due to an aging population and expanding treatment indications for chronic diseases. Simultaneously, adverse drug events-harmful and unintended events related to medication use or misuse-have increased. In Canada, adverse events to outpatient medications cause over two million emergency department visits and 700,000 hospital admissions, costing over $1 billion in healthcare expenditures annually. Optimizing the benefits of medications while limiting their potential for harm is a public health priority across patient populations, health settings and medical disciplines.

Patients with adverse drug events often seek care in hospitals due to the unexpected and serious nature of these events. After assessment and treatment, patients are discharged back into the care of a community-based provider who often cannot access the hospital's medical record, may not receive a legible or detailed discharge summary, and is at risk of either re-starting the culprit medication for chronic disease management in the case of an adverse drug reaction. The investigators developed ActionADE to address this type of information discontinuity. ActionADE was integrated to a province-wide network that links all pharmacies in British Columbia to a central data system, allowing users to see their patient's medication dispensing history.

The investigators will conduct a triple-blind randomized controlled trial to evaluate the effectiveness of ActionADE on preventing subsequent adverse drug reactions. The trial will take place in two urban tertiary care (Vancouver General and Saint Paul's Hospitals) and one urban community hospital (Lions Gate Hospital) within the Greater Vancouver area, in British Columbia, Canada. Other hospitals may be added to accelerate recruitment into the trial if approved by the British Columbia Ministry of Health.

The primary objective of the main trial is to evaluate the effect of providing information continuity about adverse drug reactions using ActionADE on culprit drug re-dispensations over 12 months compared to standard care. Secondary objectives are to evaluate the effect on outpatient and emergency department visits, admissions, hospital-days and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 years of age or older presenting to the participating emergency departments with an adverse drug reaction to a prescribed outpatient medication that was reported in ActionADE.

Exclusion Criteria:

* Patients whose adverse drug event is categorized as life threatening will be excluded.
* Patients without a Provincial Health Number will be excluded as this will prevent linkage with PharmaNet and other administrative data for outcomes ascertainment.
* Patients diagnosed with adverse drug events to culprit medications not on the provincial formulary will be excluded as we will not be able to ascertain re-dispensations outcomes for these medications using PharmaNet data.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Culprit or same-class medication re-dispensing during follow-up | 12 months
  The summary measure will be the proportion of patients with a culprit medication re-dispensation within 12 months. The effect measure will be the between-group difference in the proportion with a 12 month re-dispensation.

SECONDARY OUTCOMES:
Hospital visits | 12 months
  Number of outpatient and emergency visits
Hospital stay | 12 months
  Number of hospital-days during hospital admissions.
Mortality | 12 months
  Number of all cause mortality during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne M Hohl, MD, MSc, Principal Investigator — University of British Columbia

REFERENCES:
- [Derived] Hau JP, Brasher PMA, Cragg A, Small S, Wickham M, Hohl CM. Using ActionADE to create information continuity to reduce re-exposures to harmful medications: study protocol for a randomized controlled trial. Trials. 2021 Feb 5;22(1):119. doi: 10.1186/s13063-021-05061-7. PMID 33546752